CLINICAL TRIAL: NCT06231537
Title: Visual Oral Examination in Primary Health Care for Early Detection of Oral Cancer: Targeting High-Risk Individuals in the Municipality of Rio de Janeiro
Brief Title: Visual Oral Examination for Early Detection of Oral Cancer in High-Risk Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Marcia Frias Pinto Marinho, Principal Investigator, Ph.D. Candidate in Dentistry, Department of Oral Diagnosis and Pathology, School of Dentistry, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: O/OC 2023-2024
Record Dates: First submitted 2024-01-12; First posted 2024-01-30 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Mouth Neoplasms
Keywords: Mouth Neoplasms; early diagnosis; public health; prevention
MeSH Terms: conditions — Mouth Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Health professionals, including dentists (CD), dental hygienists (TSB), dental assistants (ASB), nurses, and general practitioners, will continue providing care to users in accordance with the existing Service Card protocols in the city of Rio de Janeiro. This ensures on-demand service for users seeking dental care. Additionally, they will continue to facilitate participation in the Tobacco Control Program for interested individuals, following the established protocol of the city of Rio de Janeiro. Notably, members of the control group will not partake in the qualification process conducted by this research project. However, in the event of positive results at the research's conclusion, consideration will be given to extending qualification opportunities to the control group as well.
- Active Screening Group (Experimental): Health professionals (Community Health Agents, dentists, dental hygienists, dental assistants, nurses, and general practitioners) will undergo training focused on preventing OC, considering risk factors and highlighting the significance of preventive oral examinations for early diagnosis. Dentist and general practitioners will receive training to conduct oral examinations, enabling them to identify suspicious lesions and potentially malignant disorders. The qualification process will be conducted through face-to-face meetings and/or videoconferencing, supplemented by educational material delivered via the widely used messaging application (WhatsApp).
  Following qualification, tobacco users and excessive alcohol users will be invited to visit the Family Clinic for oral preventive examination. After six months, in the event that a user does not attend the Family Clinic, the Health Team will conduct an active search, through home visits or community outreach in bars.
  Interventions: Diagnostic Test: Visual oral examination
- Campaign Group (Experimental): Health professionals (Community Health Agents, dentists, dental hygienists, dental assistants, nurses, and general practitioners) will be training focused on preventing OC, risk factors and highlighting the significance of preventive oral examinations for early diagnosis. Dentist and general practitioners will receive training to conduct oral examinations, enabling them to identify suspicious lesions and potentially malignant disorders. The qualification process will be conducted through face-to-face meetings or videoconferencing.
  Following qualification, tobacco and excessive alcohol users will be invited to visit the Family Clinic for oral examination. After six months, a public awareness campaign, over one month, will be conducted in the Family Clinics. This campaign will provide guidance on risk factors, signs and symptoms, and the importance of oral examinations.
  Interventions: Diagnostic Test: Visual oral examination

INTERVENTIONS:
Diagnostic Test: Visual oral examination — Oral preventive examinations in the three groups will be conducted over a one-year period. Individuals with oral injuries will be referred to stomatology, aligning with the existing protocol. Histopathological examinations of the biopsied lesions will be performed at the Oral Pathology Laboratory of the Faculty of Dentistry at the Federal University of Rio de Janeiro, following the established procedures.
  Users diagnosed with malignancy will be directed to receive treatment at the reference hospital, with monitoring carried out by the Basic Health Unit responsible for coordinating care, in accordance with the current protocol.
  In addition to histopathological examinations, the Faculty of Dentistry will be available to conduct a physical examination and biopsy if the user is not attended to by the Municipal Health Department. This additional resource ensures comprehensive care for individuals who may not have immediate access to municipal health services.
  Arms: Active Screening Group; Campaign Group

SUMMARY:
Oral cancer (OC) is a public health problem in Brazil, with high morbidity and mortality, mainly associated with late diagnosis, which implies high-cost treatments and great social impact, with aesthetic and functional sequelae. Smokers and alcoholics are at increased risk for the disease, being early detection the most effective way to increase survival. In Brazil, cancer plan recommends early diagnosis of OC through opportunistic examination, which is carried out during regular visits to the dentist. However, this strategy has not yet been able to reverse the late diagnosis, which may be due to the low access to dental appointments by the most vulnerable groups. Studies point to the effectiveness of the preventive physical examination of the mouth for early detection when directed to the high-risk population. The aim of the present study is to compare different strategies aimed at expanding the access of the high-risk population to preventive physical examination of the mouth. A cluster-randomized trial (control group and experimental groups I and II) will be carried out in Primary Health Care units in Programmatic Area 5.2 of the city of Rio de Janeiro (eight neighborhoods in the West Zone).

In the control group, there will be no change in current care. In both experimental groups, Community Agents and health professionals will be trained in OC prevention and instructed to call the users with high-risk for OC to the preventive examination of the mouth at the health unit. After 6 months, in experimental group I, an active search will be carried out for users who did not show up for the preventive examination, while in experimental group II, a campaign on OC will be carried out for a month, inviting the population to the preventive examination. After one year, the number of people at increased risk for OC examined in each group will be compared and correlated with sociodemographic and clinicopathological variables.

DETAILED DESCRIPTION:
Oral cancer (OC) is a significant public health concern in Brazil, with the country having the highest incidence of the disease in Latin America. It ranks as the fourth most common cancer among men in the southeast region. This condition carries substantial morbidity and mortality, largely due to the majority of patients being diagnosed at advanced stages, leading to elevated treatment costs, prolonged rehabilitation, and profound social impacts such as loss of labor capacity and exclusion from social environments.

Squamous cell carcinoma, constituting 90 to 95% of OC cases, primarily affects men over 50 years old, with an emerging incidence in individuals under 40. In Brazil, the lateral border of the tongue is the primary site, characterized by invasive growth, significant recurrence rates, and metastasis to regional lymph nodes.

The main etiological factors for OC include tobacco and alcohol for intraoral lesions, prolonged exposure to ultraviolet (UV) radiation for lip cancer, and, for oropharyngeal cancer, human papillomavirus (HPV) infection. Cultural characteristics, socioeconomic level, and access to public health services also contribute to the variation in oral cancer incidence.

Primary prevention is paramount and involves educating individuals on behavioral risk factors, limiting tobacco and alcohol use, sun protection for the lips, HPV vaccination for oropharyngeal cancer prevention, and maintaining a healthy diet. Secondary prevention focuses on early disease through detection for pre-clinical signs and early diagnosis for individuals exhibiting suspected symptoms.

The justification for implementing a population screening program as a public health policy is based on established criteria. While OC meets ten out of the 19 criteria presented at the Global Oral Cancer Forum in 2016, its cost-effectiveness remains unproven, unlike breast and cervical cancer, which have well-defined population screening protocols.

Although a clinical trial in Kerala, India, did not demonstrate reduced OC mortality through population monitoring, a reanalysis in 2021 highlighted the effectiveness of targeted preventive mouth examinations by trained health professionals for at-risk populations.

In many countries, including Brazil, opportunistic examinations of the mouth's soft tissues are recommended for early diagnosis of lesions, but the majority of oral cancer cases are still diagnosed at advanced stages. The National Oral Health Policy, established in 2004, aims to promote, prevent, recover, and maintain oral health through primary care and specialized dental centers.

Recognizing structural and social determinants is crucial for effective prevention, detection, and management of OC. The "inverse screening law" highlights challenges in opportunistic examinations, and barriers to accessibility and diagnostic delays persist, especially among the elderly.

Despite the current strategy in Brazil relying on opportunistic testing, the majority of OC cases are diagnosed late. Weaknesses in the city of Rio de Janeiro, including low population coverage in Oral Health in Primary Care and limited access for at-risk populations, underscore the likely ineffectiveness of the current preventive strategy.

The present study is justified by the imperative to expand access to preventive oral examinations for individuals at increased risk for OC, aiming for early diagnosis and subsequently reducing mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are regular smokers and/or chronic alcohol users
* Individuals registered as patients at Family Clinics within Programmatic Area 5.2 in the city of Rio de Janeiro
* Individuals aged 35 years or older

Exclusion Criteria:

* Individuals who have had a regular dental visit within the last 12 months

Ages: 35 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1152 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Preventive Oral Examinations among Individuals Aged 35 and Older, Smokers, and/or Alcohol Drinkers within One Year Post-Implementation of Strategies in Experimental Groups | one year
  The descriptive characterization of the sample will be estimated for both the control and experimental groups, encompassing the absolute and relative counts of individuals aged 35 and older, smokers, and/or alcohol drinkers who underwent a preventive oral examination within one year following the implementation of strategies in the experimental groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Units of the Municipality of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutkowska M, Hnitecka S, Nahajowski M, Dominiak M, Gerber H. Oral cancer: The first symptoms and reasons for delaying correct diagnosis and appropriate treatment. Adv Clin Exp Med. 2020 Jun;29(6):735-743. doi: 10.17219/acem/116753. PMID 32598579
- [Background] Gormley M, Gray E, Richards C, Gormley A, Richmond RC, Vincent EE, Dudding T, Ness AR, Thomas SJ. An update on oral cavity cancer: epidemiological trends, prevention strategies and novel approaches in diagnosis and prognosis. Community Dent Health. 2022 Aug 30;39(3):197-205. doi: 10.1922/CDH_00032Gormley09. PMID 35852216
- [Background] Walsh T, Warnakulasuriya S, Lingen MW, Kerr AR, Ogden GR, Glenny AM, Macey R. Clinical assessment for the detection of oral cavity cancer and potentially malignant disorders in apparently healthy adults. Cochrane Database Syst Rev. 2021 Dec 10;12(12):CD010173. doi: 10.1002/14651858.CD010173.pub3. PMID 34891214
- [Background] Hertrampf K, Jurgensen M, Wahl S, Baumann E, Wenz HJ, Wiltfang J, Waldmann A. Early detection of oral cancer: a key role for dentists? J Cancer Res Clin Oncol. 2022 Jun;148(6):1375-1387. doi: 10.1007/s00432-022-03962-x. Epub 2022 Mar 6. PMID 35249159
- [Background] Zamani M, Gronhoj C, Jensen DH, Carlander AF, Agander T, Kiss K, Olsen C, Baandrup L, Nielsen FC, Andersen E, Friborg J, von Buchwald C. The current epidemic of HPV-associated oropharyngeal cancer: An 18-year Danish population-based study with 2,169 patients. Eur J Cancer. 2020 Jul;134:52-59. doi: 10.1016/j.ejca.2020.04.027. Epub 2020 May 24. PMID 32460181
- [Background] Nielsen KJ, Jakobsen KK, Jensen JS, Gronhoj C, Von Buchwald C. The Effect of Prophylactic HPV Vaccines on Oral and Oropharyngeal HPV Infection-A Systematic Review. Viruses. 2021 Jul 11;13(7):1339. doi: 10.3390/v13071339. PMID 34372545
- [Background] Abati S, Bramati C, Bondi S, Lissoni A, Trimarchi M. Oral Cancer and Precancer: A Narrative Review on the Relevance of Early Diagnosis. Int J Environ Res Public Health. 2020 Dec 8;17(24):9160. doi: 10.3390/ijerph17249160. PMID 33302498
- [Background] Nagao T, Warnakulasuriya S. Screening for oral cancer: Future prospects, research and policy development for Asia. Oral Oncol. 2020 Jun;105:104632. doi: 10.1016/j.oraloncology.2020.104632. Epub 2020 Apr 18. PMID 32315954
- [Background] Thankappan K, Subramanian S, Balasubramanian D, Kuriakose MA, Sankaranarayanan R, Iyer S. Cost-effectiveness of oral cancer screening approaches by visual examination: Systematic review. Head Neck. 2021 Nov;43(11):3646-3661. doi: 10.1002/hed.26816. Epub 2021 Jul 14. PMID 34260118
- [Background] Cheung LC, Ramadas K, Muwonge R, Katki HA, Thomas G, Graubard BI, Basu P, Sankaranarayanan R, Somanathan T, Chaturvedi AK. Risk-Based Selection of Individuals for Oral Cancer Screening. J Clin Oncol. 2021 Feb 20;39(6):663-674. doi: 10.1200/JCO.20.02855. Epub 2021 Jan 15. PMID 33449824
- [Background] Sankaranarayanan R, Ramadas K, Thara S, Muwonge R, Thomas G, Anju G, Mathew B. Long term effect of visual screening on oral cancer incidence and mortality in a randomized trial in Kerala, India. Oral Oncol. 2013 Apr;49(4):314-21. doi: 10.1016/j.oraloncology.2012.11.004. Epub 2012 Dec 21. PMID 23265945
- [Background] Bouvard V, Nethan ST, Singh D, Warnakulasuriya S, Mehrotra R, Chaturvedi AK, Chen TH, Ayo-Yusuf OA, Gupta PC, Kerr AR, Tilakaratne WM, Anantharaman D, Conway DI, Gillenwater A, Johnson NW, Kowalski LP, Leon ME, Mandrik O, Nagao T, Prasad VM, Ramadas K, Roitberg F, Saintigny P, Sankaranarayanan R, Santos-Silva AR, Sinha DN, Vatanasapt P, Zain RB, Lauby-Secretan B. IARC Perspective on Oral Cancer Prevention. N Engl J Med. 2022 Nov 24;387(21):1999-2005. doi: 10.1056/NEJMsr2210097. Epub 2022 Oct 18. No abstract available. PMID 36378601
- [Background] Bouvard V, Wentzensen N, Mackie A, Berkhof J, Brotherton J, Giorgi-Rossi P, Kupets R, Smith R, Arrossi S, Bendahhou K, Canfell K, Chirenje ZM, Chung MH, Del Pino M, de Sanjose S, Elfstrom M, Franco EL, Hamashima C, Hamers FF, Herrington CS, Murillo R, Sangrajrang S, Sankaranarayanan R, Saraiya M, Schiffman M, Zhao F, Arbyn M, Prendiville W, Indave Ruiz BI, Mosquera-Metcalfe I, Lauby-Secretan B. The IARC Perspective on Cervical Cancer Screening. N Engl J Med. 2021 Nov 11;385(20):1908-1918. doi: 10.1056/NEJMsr2030640. No abstract available. PMID 34758259
- [Background] Ribeiro MFA, Oliveira MCM, Leite AC, Bruzinga FFB, Mendes PA, Grossmann SMC, de Araujo VE, Souto GR. Assessment of screening programs as a strategy for early detection of oral cancer: a systematic review. Oral Oncol. 2022 Jul;130:105936. doi: 10.1016/j.oraloncology.2022.105936. Epub 2022 Jun 2. PMID 35662028
- [Background] D'souza S, Addepalli V. Preventive measures in oral cancer: An overview. Biomed Pharmacother. 2018 Nov;107:72-80. doi: 10.1016/j.biopha.2018.07.114. Epub 2018 Aug 3. PMID 30081204
- [Background] Carlander AF, Jakobsen KK, Bendtsen SK, Garset-Zamani M, Lynggaard CD, Jensen JS, Gronhoj C, Buchwald CV. A Contemporary Systematic Review on Repartition of HPV-Positivity in Oropharyngeal Cancer Worldwide. Viruses. 2021 Jul 9;13(7):1326. doi: 10.3390/v13071326. PMID 34372532
- [Background] Bosetti C, Carioli G, Santucci C, Bertuccio P, Gallus S, Garavello W, Negri E, La Vecchia C. Global trends in oral and pharyngeal cancer incidence and mortality. Int J Cancer. 2020 Aug 15;147(4):1040-1049. doi: 10.1002/ijc.32871. Epub 2020 Jan 30. PMID 31953840
- [Background] Chaturvedi AK, Anderson WF, Lortet-Tieulent J, Curado MP, Ferlay J, Franceschi S, Rosenberg PS, Bray F, Gillison ML. Worldwide trends in incidence rates for oral cavity and oropharyngeal cancers. J Clin Oncol. 2013 Dec 20;31(36):4550-9. doi: 10.1200/JCO.2013.50.3870. Epub 2013 Nov 18. PMID 24248688
- [Background] Sallam M, Dababseh D, Yaseen A, Al-Haidar A, Ettarras H, Jaafreh D, Hasan H, Al-Salahat K, Al-Fraihat E, Hassona Y, Sahin GO, Mahafzah A. Lack of knowledge regarding HPV and its relation to oropharyngeal cancer among medical students. Cancer Rep (Hoboken). 2022 Jul;5(7):e1517. doi: 10.1002/cnr2.1517. Epub 2021 Jul 22. PMID 34291614
- [Background] Gupta AK, Kanaan M, Siddiqi K, Sinha DN, Mehrotra R. Oral Cancer Risk Assessment for Different Types of Smokeless Tobacco Products Sold Worldwide: A Review of Reviews and Meta-analyses. Cancer Prev Res (Phila). 2022 Nov 1;15(11):733-746. doi: 10.1158/1940-6207.CAPR-21-0567. PMID 36095092
- [Background] Saxena R, Prasoodanan P K V, Gupta SV, Gupta S, Waiker P, Samaiya A, Sharma AK, Sharma VK. Assessing the Effect of Smokeless Tobacco Consumption on Oral Microbiome in Healthy and Oral Cancer Patients. Front Cell Infect Microbiol. 2022 Mar 31;12:841465. doi: 10.3389/fcimb.2022.841465. eCollection 2022. PMID 35433507
- [Background] Warnakulasuriya S. Global epidemiology of oral and oropharyngeal cancer. Oral Oncol. 2009 Apr-May;45(4-5):309-16. doi: 10.1016/j.oraloncology.2008.06.002. Epub 2008 Sep 18. PMID 18804401
- [Background] Du M, Nair R, Jamieson L, Liu Z, Bi P. Incidence Trends of Lip, Oral Cavity, and Pharyngeal Cancers: Global Burden of Disease 1990-2017. J Dent Res. 2020 Feb;99(2):143-151. doi: 10.1177/0022034519894963. Epub 2019 Dec 24. PMID 31874128
- [Background] O'Connor R, Schneller LM, Felicione NJ, Talhout R, Goniewicz ML, Ashley DL. Evolution of tobacco products: recent history and future directions. Tob Control. 2022 Mar;31(2):175-182. doi: 10.1136/tobaccocontrol-2021-056544. PMID 35241585
- [Background] Sultan AS, Jessri M, Farah CS. Electronic nicotine delivery systems: Oral health implications and oral cancer risk. J Oral Pathol Med. 2021 Mar;50(3):316-322. doi: 10.1111/jop.12810. Epub 2018 Dec 14. PMID 30507043
- [Background] Wilson C, Tellez Freitas CM, Awan KH, Ajdaharian J, Geiler J, Thirucenthilvelan P. Adverse effects of E-cigarettes on head, neck, and oral cells: A systematic review. J Oral Pathol Med. 2022 Feb;51(2):113-125. doi: 10.1111/jop.13273. PMID 35048431
- [Background] Dal Maso L, Torelli N, Biancotto E, Di Maso M, Gini A, Franchin G, Levi F, La Vecchia C, Serraino D, Polesel J. Combined effect of tobacco smoking and alcohol drinking in the risk of head and neck cancers: a re-analysis of case-control studies using bi-dimensional spline models. Eur J Epidemiol. 2016 Apr;31(4):385-93. doi: 10.1007/s10654-015-0028-3. Epub 2015 Apr 9. PMID 25855002
- [Background] LeHew CW, Weatherspoon DJ, Peterson CE, Goben A, Reitmajer K, Sroussi H, Kaste LM. The Health System and Policy Implications of Changing Epidemiology for Oral Cavity and Oropharyngeal Cancers in the United States From 1995 to 2016. Epidemiol Rev. 2017 Jan 1;39(1):132-147. doi: 10.1093/epirev/mxw001. PMID 28402398
- [Background] Ahuja NA, Kedia SK, Ward KD, Pichon LC, Chen W, Dillon PJ, Navaparia H. Effectiveness of Interventions to Improve Oral Cancer Knowledge: a Systematic Review. J Cancer Educ. 2022 Jun;37(3):479-498. doi: 10.1007/s13187-021-01963-x. Epub 2021 Jan 27. PMID 33506408
- [Background] Shaffer KM, Turner KL, Siwik C, Gonzalez BD, Upasani R, Glazer JV, Ferguson RJ, Joshua C, Low CA. Digital health and telehealth in cancer care: a scoping review of reviews. Lancet Digit Health. 2023 May;5(5):e316-e327. doi: 10.1016/S2589-7500(23)00049-3. PMID 37100545
- [Background] Warnakulasuriya S, Kerr AR. Oral Cancer Screening: Past, Present, and Future. J Dent Res. 2021 Nov;100(12):1313-1320. doi: 10.1177/00220345211014795. Epub 2021 May 26. PMID 34036828
- [Background] Warnakulasuriya S. Oral potentially malignant disorders: A comprehensive review on clinical aspects and management. Oral Oncol. 2020 Mar;102:104550. doi: 10.1016/j.oraloncology.2019.104550. Epub 2020 Jan 22. PMID 31981993
- [Background] Mandrik O, Roitberg F, Lauby-Secretan B, Parak U, Ramadas K, Varenne B, Sankaranarayanan R, Carvalho AL. Perspective on oral cancer screening: Time for implementation research and beyond. J Cancer Policy. 2023 Mar;35:100381. doi: 10.1016/j.jcpo.2022.100381. Epub 2023 Jan 2. PMID 36599217
- [Background] Netuveli G, Sheiham A, Watt RG. Does the 'inverse screening law' apply to oral cancer screening and regular dental check-ups? J Med Screen. 2006;13(1):47-50. doi: 10.1258/096914106776179836. PMID 16569306
- [Background] Sankaranarayanan R, Ramadas K, Thomas G, Muwonge R, Thara S, Mathew B, Rajan B; Trivandrum Oral Cancer Screening Study Group. Effect of screening on oral cancer mortality in Kerala, India: a cluster-randomised controlled trial. Lancet. 2005 Jun 4-10;365(9475):1927-33. doi: 10.1016/S0140-6736(05)66658-5. PMID 15936419
- [Background] Scott SE, Rizvi K, Grunfeld EA, McGurk M. Pilot study to estimate the accuracy of mouth self-examination in an at-risk group. Head Neck. 2010 Oct;32(10):1393-401. doi: 10.1002/hed.21341. PMID 20146330